CLINICAL TRIAL: NCT06081231
Title: The Safety and Efficacy of Open-Source Artificial Pancreas System Among People With Type 1 Diabetes Mellitus in China
Brief Title: Open-Source Artificial Pancreas System Use Among People With Type 1 Diabetes Mellitus in China
Status: Recruiting | Type: Observational
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jinhua Yan, Vice Professor,Principal Investigator,Department of Endocrinology and Metabolism, Third Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: MLei2
Record Dates: First submitted 2023-09-26; First posted 2023-10-13 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: artificial pancreas system; automated insulin delivery; do-it-yourself; closed loop; open source
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- open-source APS: open-source APS consisted of an insulin pump, a CGM system, and a heuristic algorithm on an Android smartphone.
  Interventions: Device: open-source APS;

INTERVENTIONS:
Device: open-source APS; — a continuous glucose monitoring system, an insulin pump, and an intelligent algorithm.

SUMMARY:
This real-world observational study aims to reveal the current status of the open-source artificial pancreas system (APS) use among people with T1DM in China and assess the glycemic efficacy and potential related factors of the open-source APS.

DETAILED DESCRIPTION:
This is a real-world observational study analyzing data on open-source artificial pancreas systems(APS) in people with T1DM in China. Data will collected during clinical routine, questionnaires, standard-of-care laboratory tests, and CGM data among whom are willing to share. Baseline data from before the start (up to -3 months) of the open-source APS system and follow-up data at 3, 6, 9, 12, and the following period will be analyzed when available. There are no medical interventions, extra visits, or laboratory tests planned outside the normal clinical routine. Glycemic control and patient-reported outcomes during follow-up will be compared with glycemic control and patient-reported outcome data at baseline.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed T1DM.
2. Currently use open-source APS for at least 3 months.
3. Willing and able to provide informed consent (or be a parent or other legally authorized representative) and to provide the data.
4. reside in China.

Exclusion Criteria:

None

Ages: 3 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: people with T1DM regardless of age or pregnant state.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
proportion of time spent in the target glucose range | baseline(at least 2 weeks before the start of APS), and 3 months,6 months, 9 months, 12 months, and following period after the start of APS
  time in range(TIR, 70-180mg/dL)

SECONDARY OUTCOMES:
proportion of time spent in the hypoglycemic range | baseline(at least 2 weeks before the start of APS), and 3 months,6 months, 9 months, 12 months, and following period after the start of APS
  time below range(TBR, <70mg/dL;<54mg/dL)
proportion of time spent in the hyperglycemic range | baseline(at least 2 weeks before the start of APS), and 3 months,6 months, 9 months, 12 months, and following period after the start of APS
  time above range(TAR, >180mg/dL;>250mg/dL)
concentration of HbA1c | baseline(at least 2 weeks before the start of APS), and 3 months,6 months, 9 months, 12 months, and following period after the start of APS
  glycated hemoglobin A1C

CONTACTS AND LOCATIONS:
Overall Officials: Jinhua Yan, PHD,MD, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Jinhua Yan, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No